CLINICAL TRIAL: NCT02559076
Title: Preschool Obesity in the United Arab Emirates: Determinants and the Effectiveness of the 10-step Healthy Lifestyle Tool for Toddlers- Eat Right Emirates
Brief Title: The Eat Right Emirates Healthy Lifestyle Study
Acronym: ERERCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Collaborators: United Arab Emirates University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 14NT05
Record Dates: First submitted 2015-09-11; First posted 2015-09-24 (Estimated); Last update posted 2015-09-25 (Estimated); Status verified 2015-09

CONDITIONS: Childhood Obesity; Dietary Habits
Keywords: Overweight; Obesity; Preschool children; United Arab Emirates; Dietary patterns; BMI z-scores
MeSH Terms: conditions — Pediatric Obesity; Feeding Behavior; Overweight; Obesity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ten Steps Leaflet (Experimental): Ten steps leaflet advice for healthy lifestyle
  Interventions: Behavioral: Ten Steps leaflet advice for healthy lifestyle
- Usual care (No Intervention): Usual care given

INTERVENTIONS:
Behavioral: Ten Steps leaflet advice for healthy lifestyle — Ten steps leaflet advice for healthy lifestyle
  Arms: Ten Steps Leaflet

SUMMARY:
The aim of the present study was to investigate the potential factors that determine preschool obesity in Al Ain, United Arab Emirates, and assess the effectiveness of a simple healthy lifestyle tool: Eat Right Emirates (ERE) adapted from the Ten Steps for Healthy Toddlers, produced in the UK by the Infant and Toddler Forum.

DETAILED DESCRIPTION:
Study Aims

The aim of this study is to identify social, developmental and dietary risk factors, which predispose to obesity in preschool Emirati children and to assess the effectiveness of a simple healthy lifestyle tool: Eat Right Emirates (ERE) adapted from the Ten Steps for Healthy Toddlers, produced in the UK by the Infant and Toddler Forum using an RCT study design.

Primary Research Questions

1. Do dietary patterns influence obesity risk in Emirati children aged 3-4 years?
2. Are dietary and other behaviours associated with obesity risk in Kuwaiti preschool children?
3. Are developmental factors, associated with obesity risk in Emirati preschool children?

Secondary Research Questions

1. Does a healthy lifestyle intervention improve eating behaviour and physical activity in Emirati preschool children?

Investigation Plan

Determinants of obesity in children aged 3-4 years attending preschool centres in UAE will be investigated within a cross-sectional observation study. Dietary intake will be assessed using food records and questionnaires. These will be analysed to give information on dietary patterns and nutritional intake. Developmental factors, such as infant feeding and growth patterns and other lifestyle behaviours that may influence obesity risk, such as physical activity and food related behaviours, will also be evaluated using questionnaires. Obesity will be assessed using non-invasive methods to measure body size and fatness. Risk factors for CVD including blood pressure and pulse wave velocity will also be assessed using non-invasive methods.

The same infants and mothers will be followed-up one year later to allow:

1. Investigation into tracking of risk factors in preschool children.
2. Study of the impact of risk factors on change in BMI during the preschool period.

The cohort will then provide a resource to investigate the determinants of obesity in preschool children from UAE.

Recruitment

The study population of preschool children will be recruited from an existing sub-sample of parents who took part in a previous study in Al Ain district, Abu Dhabi. The study population will therefore be representative of the general Emirati population. Parents will be contacted prior to the study, with permission from the Ministry of Health.

Data collection

The potential determinants of obesity in preschool Emirati children (exposures) and effects on obesity and risk factors for CVD (outcomes) will be investigated as detailed below. Data will be collected at baseline and at follow up one year later. All measurements will be undertaken by trained team members and performed according to the UCL CNRC standard operational procedures.

All testing procedures will take place on the school premises with parents present.

Exposures

Exposures investigated in this study include growth patterns, infant/child feeding practices, dietary patterns, appetite characteristics and dietary behaviours .

Dietary Patterns and Intake

Dietary patterns in mothers and children will be assessed using a food frequency questionnaire (FFQ). Mothers will also be asked to complete a 5-day food diary representative of their child's usual diet at study baseline and one-year follow up. Diaries will be analysed for all nutrients with UK dietary reference values using dietary analysis software based on food composition data from the 6th edition of McCance and Widdowson's composition of foods.

Medical History and Sociodemographic Factors

Information on child and parental sociodemographic characteristics and medical history will be collected using questionnaires. Parental anthropometry will be measured where possible to give a measure of genetic exposures.

Lifestyle Practices

Parental and child diet will be assessed using validated questionnaires.

Outcome measures:

Anthropometry Cardiovascular health

ELIGIBILITY:
Inclusion Criteria:

* Healthy preschool children

Exclusion Criteria:

* Pre-existing medical condition
* Physical disability
* Social problems

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2014-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Dietary patterns will be assessed using a food frequency questionnaire (FFQ). | 6 months
  Dietary Patterns will be compared between randomized groups following intervention.

SECONDARY OUTCOMES:
Body Mass Index | 6 months
  Body mass index (weight (kg)/height(m2) will be compared between randomized groups following intervention.